CLINICAL TRIAL: NCT02904655
Title: Dietary Interventions in Asthma Treatment:Healthy Eating Better Breathing Asthma Diet Pilot Study
Brief Title: Healthy Eating Better Breathing: A Feeding Study in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NA_00071879
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy diet (Active Comparator): Participants were provided all meals and snacks for four weeks. Menus were created to target a healthy diet high in unsaturated fats.
  Interventions: Other: healthy diet
- control diet (No Intervention): Participants were instructed to consume their usual diet.

INTERVENTIONS:
Other: healthy diet — Participants were provided meals and snacks for one month that represented a healthy diet that is high in unsaturated fats, approximating a Mediterranean diet
  Arms: healthy diet

SUMMARY:
The study is a randomized, crossover meal-replacement pilot intervention to determine feasibility of a larger scale dietary trial in asthma and gather preliminary evidence for the impact of a healthy diet on asthma outcomes. Participants with doctor-diagnosed asthma were randomized to crossover trial of a 4-week dietary intervention or usual diet with a 4-week washout period. During the dietary intervention, all meals and snacks were provided by the study.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate feasibility of a randomized, controlled clinical trial of a dietary intervention in a population of adults with asthma and to determine sample size estimates for a larger, more definitive trial aimed at improving asthma clinical outcomes and improving markers of inflammation and oxidative stress. The study uses a feeding trial design comprised of a 4 week dietary intervention in which all meals are provided to study participants and a 4 week control diet comprised of usual dietary intake. Participants are randomized to the intervention or control diet and then cross over to the alternate assignment after a 4 week washout period.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-50, self-reported physician diagnosis and treatment for asthma within the 12 months prior to enrollment, stable asthma defined as no asthma exacerbation (emergency department visit, systemic steroid treatment, or urgent care visit) or respiratory infection in the 4 weeks prior to enrollment.

Exclusion Criteria:

* active smokers,pregnant or breastfeeding, using systemic corticosteroids or warfarin, had another major pulmonary diagnosis or significant systemic illness, reported excessive alcohol consumption (over 14 drinks per week or six or more drinks on one or more occasions per week), reported food allergy, or weighed over 350 pounds or changed weight by over ten pounds in the two months prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participant drop outs | Change from baseline and 4 weeks
  Feasibility will be assessed by the number of drop outs.
Adherence using 24 hour diet recall | Change from baseline to 4 weeks
  Adherence to the dietary intervention will be assessed using self-report of dietary intake via 24 hour dietary recall.
Adherence assessed by serum carotenoids | Change from baseline to 4 weeks
  Serum carotenoids will be measured at baseline and at 4 weeks. An increase in serum carotenoids is expected with adherence to the dietary intervention.

SECONDARY OUTCOMES:
FEV1 | Difference between baseline and 4 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1) will be assessed and compared between baseline and 4 weeks after the dietary intervention
FEV1 | Difference between baseline and 2 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1) will be assessed and compared between baseline and 2 weeks after the dietary intervention
FVC | Difference between baseline and 2 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced vital capacity (FVC) will be assessed and compared between baseline and 4 weeks after the dietary intervention
FVC | Difference between baseline and 4 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced vital capacity (FVC) will be assessed and compared between baseline and 4 weeks after the dietary intervention
FEV1/FVC ratio | Difference between baseline and 4 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio will be assessed and compared between baseline and 4 weeks after the dietary intervention
FEV1/FVC ratio | Difference between baseline and 2 weeks
  Spirometry will be measured according to the American Thoracic Society standards. The forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio will be assessed and compared between baseline and 2 weeks after the dietary intervention
Asthma status | Difference between baseline and 4 weeks
  Asthma Control Test (ACT, range 5-25, higher score denoting better asthma control). The change in score between baseline and week 4 will be assessed.
Asthma status | Difference between baseline and 2 weeks
  Asthma Control Test (ACT, range 5-25, higher score denoting better asthma control). The change in score between baseline and week 2 will be assessed.
Asthma Symptom Utility Index | Difference between baseline and 4 weeks
  Asthma Symptom Utility Index (ASUI, range 0-1, higher score denoting fewer symptoms) will be measured and the difference between week 4 and week 0 will be assessed.
Asthma Symptom Utility Index | Difference between baseline and 2 weeks
  Asthma Symptom Utility Index (ASUI, range 0-1, higher score denoting fewer symptoms) will be measured and the difference between week 2 and week 0 (baseline) will be assessed.
Asthma Quality of Life Questionnaire (AQLQ) | Difference between baseline and 4 weeks
  Asthma Quality of Life Questionnaire (AQLQ) is a 32 item questionnaire and each question uses a 7-point Likert scale (7 = not impaired at all; - 1 = severely impaired). Scores between week 0 (baseline) and week 4 will be assessed.
Asthma Quality of Life Questionnaire (AQLQ) | Difference between baseline and 2 weeks
  Asthma Quality of Life Questionnaire (AQLQ) is a 32 item questionnaire and each question uses a 7-point Likert scale (7 = not impaired at all - 1 = severely impaired). Scores between week 0 (baseline) and week 2 will be assessed.
Exhaled nitric oxide | Difference between baseline and 4 weeks
  Exhaled nitric oxide is an indicator of airway inflammation and will be measured according to American Thoracic Society standards at baseline and 4 weeks.
Exhaled nitric oxide | Difference between baseline and 2 weeks
  Exhaled nitric oxide is an indicator of airway inflammation and will be measured according to American Thoracic Society standards at baseline and 2 weeks.
Adherence assessed by serum carotenoids | Difference between baseline and 2 weeks
  Serum carotenoids will be measured at baseline and at 4 weeks. An increase in serum carotenoids is expected with adherence to the dietary intervention.

IPD SHARING:
Plan to Share IPD: No